CLINICAL TRIAL: NCT01015781
Title: Multi-Site Evaluation of Progressive Tinnitus Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C7213-R
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Tinnitus
Keywords: Tinnitus; Counseling; Education; Rehabilitation of hearing impaired; Triage; Evaluation studies; Quality of health care
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Progressive Tinnitus Management
  Interventions: Procedure: Progressive Tinnitus Management
- Arm 2 (Other): Wait List Control
  Interventions: Procedure: Wait List Control

INTERVENTIONS:
Procedure: Progressive Tinnitus Management — The program follows a five-level "progressive intervention" model that addresses the various needs of tinnitus patients in a systematic and hierarchical manner-from initial contact with a VA provider through long-term treatment. The five levels of progressive intervention are: 1) Triage; 2) Audiologic Evaluation; 3) Group Education; 4) Interdisciplinary Evaluation; 5) Individualized Support
  Other Names: PTM
  Arms: Arm 1
Procedure: Wait List Control — VA audiologists typically (a) perform an audiologic evaluation; (b) fit hearing aids if necessary; and (c) provide basic information about tinnitus in the form of one-time, one-on-one informational counseling and/or a tinnitus handout. We therefore will provide these procedures for subjects who are randomized to receive usual care. Usual care subjects also can be referred for other clinical services as deemed appropriate.
  Arms: Arm 2

SUMMARY:
This multi-site study evaluated the implementation of Progressive Tinnitus Management (PTM), which combines both Audiology and Psychology approaches to Tinnitus Management. Those Veterans who require intervention for tinnitus have different levels of need, and this progressive approach gives them the appropriate level of intervention.

DETAILED DESCRIPTION:
Objectives. We completed a single-site pilot project to develop and evaluate Progressive Tinnitus Management (PTM). PTM takes into account the fact that most Veterans who complain of tinnitus do not require extensive intervention. The method thus is "progressive" in that a hierarchical approach is used to provide clinical services only to the degree needed by individual patients. Preliminary analyses of our pilot data provide evidence that PTM is an effective and efficient means of providing tinnitus management services to Veterans. Importantly, The Veterans Affairs (VA) Audiology and Speech Pathology Program Office has identified PTM as a standardized method of tinnitus management for use at all VA medical centers. It is essential to more definitively evaluate PTM for routine application at VA medical centers. Accordingly, the specific aim of this study was to conduct a randomized clinical trial at multiple VA medical centers to evaluate the effectiveness and clinical utility of PTM as compared to Wait List Control.

Plan. The 3-year study was based at the VA National Center for Rehabilitative Auditory Research (NCRAR), and PTM was implemented and evaluated in a randomized clinical trial at the Memphis VA Medical Center and at the VA Connecticut Healthcare System (West Haven). During months 0-6: (a) All clinical materials for conducting PTM were modified (especially with the addition of Cognitive-Behavioral Therapy - CBT); (b) training materials were developed (the web-based PTM training program for VA audiologists was updated; PTM training will be developed for VA psychologists); (c) by random selection, five audiologists (two in Memphis, three in West Haven) were identified to conduct PTM and five (two in Memphis, three in West Haven) were identified to conduct usual care; (d) the five PTM audiologists (the West Haven study psychologist developed the training). By month 7, the randomized clinical trial was implemented at the two VA sites and continued through year 3.

Methods. Prior to conducting the clinical trial, PTM was modified to incorporate critical components of CBT at all levels of intervention so as to address the psychological effects of tinnitus. Qualifying Veteran subjects (n=150 at each site) were randomized into either PTM or Wait List Control. Self-perceived tinnitus handicap was evaluated pre- and post-intervention for each subject using the Tinnitus Handicap Inventory. The five audiologists and two psychologists who participate in this study were interviewed to determine their level of satisfaction with the PTM protocol to which they are assigned. Evaluation of the program will determine its efficacy, and will identify areas of needed improvement.

Relevance to VA's Mission. Although tinnitus is the second most common service-connected disability, most VA medical centers do not provide comprehensive clinical services for Veterans suffering from tinnitus. This study extends our current work, which has focused on the development of a comprehensive tinnitus management protocol that can be implemented efficiently in VA hospitals. Further development of PTM has the potential of providing needed tinnitus services to Veterans across the country for a relatively small cost and with minimal impact on individual VA hospitals.

ELIGIBILITY:
Inclusion Criteria:

* are eligible for audiology services at their respective VAMC;
* report the chronic presence of tinnitus (i.e., they have tinnitus that they can usually hear when they listen for it in a quiet room);
* report that their tinnitus is at least a "small" problem; and
* are willing to give verbal consent.

Exclusion Criteria:

* are not Veterans;
* have received previous tinnitus services at their VAMC;
* report that their tinnitus is "no problem";
* are unable (for any reason) to fulfill all of the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Henry, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (3):
- United States (3):
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Medical Center, Memphis, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Care: Immediate Care: The program follows a five-level "progressive intervention" model that addresses the various needs of tinnitus patients in a systematic and hierarchical manner-from initial contact with a VA provider through long-term treatment. The five levels of progressive intervention are: 1) Triage; 2) Audiologic Evaluation; 3) Group Education; 4) Interdisciplinary Evaluation; 5) Individualized Support
- Wait List Control: Wait List Control: VA audiologists typically (a) perform an audiologic evaluation; (b) fit hearing aids if necessary; and (c) provide basic information about tinnitus in the form of one-time, one-on-one informational counseling and/or a tinnitus handout. We therefore will provide these procedures for subjects who are randomized to receive usual care. Wait List Control subjects also can be referred for other clinical services as deemed appropriate.
Period: Overall Study
Arm/Group | Immediate Care | Wait List Control
Started | 150 | 150
Completed | 113 | 121
Not Completed | 37 | 29

BASELINE CHARACTERISTICS:
Groups:
- Immediate Care: The program follows a five-level "progressive intervention" model that addresses the various needs of tinnitus patients in a systematic and hierarchical manner-from initial contact with a VA provider through long-term treatment. The five levels of progressive intervention are: 1) Triage; 2) Audiologic Evaluation; 3) Group Education; 4) Interdisciplinary Evaluation; 5) Individualized Support
- Wait List Control: VA audiologists typically (a) perform an audiologic evaluation; (b) fit hearing aids if necessary; and (c) provide basic information about tinnitus in the form of one-time, one-on-one informational counseling and/or a tinnitus handout. We therefore will provide these procedures for subjects who are randomized to receive usual care. Wait List Control subjects also can be referred for other clinical services as deemed appropriate.
- Total: Total of all reporting groups
Arm/Group | Immediate Care | Wait List Control | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.72 (13.92) | 58.05 (12.05) | 57.89 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 145 | 141 | 286
Region of Enrollment [Number; unit: participants]
  United States | 150 | 150 | 300

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Functional Index Change Score
Description: The Tinnitus Functional Index (TFI) is a tinnitus outcome measure that has been validated for "responsiveness" (Meikle et al., 2012). Prior to the TFI, no tinnitus questionnaire had been specifically designed and tested to maximize responsiveness to treatment-related change.
  Completion of the 25-item TFI results in an index score that can range from 0 to 100, with higher scores reflecting greater problems associated with tinnitus. The following is a general guide to facilitate interpretation of TFI scores:
  * <25 = relatively mild tinnitus (little or no need for intervention)
  * 25-50 = significant problems with tinnitus (possible need for intervention) •>50 = tinnitus severe enough to qualify for more aggressive intervention Data from the TFI development study (Meikle et al., 2012) suggest that a reduction in the TFI score of at least 13 points would indicate a clinical improvement that a patient would consider important or meaningful.
Time Frame: Baseline, 6 months (from Baseline)
Population: The analysis was "intention to treat (ITT)". Includes all subjects from whom both baseline and 6 month data were collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Care | Wait List Control
Number analyzed (Participants) | 112 | 119
units on a scale | -5.71 (18.77) | .8 (17.47)

ADVERSE EVENTS:
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study
Arm/Group | Immediate Care | Wait List Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes